## A RANDOMIZED SHAM-CONTROLLED STUDY OF HOME-DELIVERED NON-INVASIVE NEUROSTIMULATION FOR MIGRAINE [IRB#19008-01, NCT03874351]

## STATISTICAL ANALYSIS PLAN

(UPDATE 1.29.20)

## **Analysis Plan (Update 1.29.20)**

Participants will be randomized within randomly selected blocks of sizes 2, 4, and 6. The randomization list will be generated by an investigator not otherwise associated with the administration of treatment or collection of data.

All patient characteristics and outcomes will be evaluated for distribution. For all bivariate tests, the appropriate parametric or non-parametric test will be selected based on distribution. Patient characteristics will be described and bivariate tests will evaluate any differences across treatment group (active tDCS vs. sham tDCS). Primary and secondary outcomes at baseline will be described and bivariate tests will evaluate any differences across group. Bivariate tests will evaluate differences in attrition, patient satisfaction, adverse events (including all adverse events, serious adverse events, and adverse events attributed to the treatment), and quality of blinding across group.

All outcomes will be described using data visualization. Differences in outcome between the active tDCS and sham tDCS groups will be evaluated in both intent-to-treat and completer analysis using non-parametric statistics as appropriate (see Table below). Intent-to-treat analysis will impute missing values using all available data. Differences in outcome between people with chronic (15 or more headache days/month) vs. episodic migraine, with and without medication overuse (e.g., using a MSM on 10 or more days per month during the baseline period), and with high and low levels of patient compliance will also be evaluated using the appropriate non-parametric statistic.

Alpha will be set at 0.05, two-tailed, for all analyses. SPSS v. 25.0 and R will be used for all analyses.

| Primary Outcome | Description | Tentative Analysis Type |
|---|---|---|
| Change in migraine day/30 | Median change in the number | Mann-Whitney U |
| day | of migraine days per 30 day | |
| | period, from M0 to M2. | |
| Secondary Outcomes | | |
| Responders | % of participants who report | Fisher's Exact Test |
| | a 50% reduction in migraine | |
| | days, from M0 to M2. | |
| Change in headache attack/30 | Median change in number of | Mann-Whitney U |
| days | attacks per 30 day period, | |
| | from M0 to M2. | |
| Change in courts medication | Madian abanga in number of | Monn Whitney II |
| Change in acute medication | Median change in number of days on which an acute | Mann-Whitney U |
| use | medication was used from | |
| | M0 to M2. | |
| Change in headache attack | Median change in NRS from | Mann-Whitney U |
| intensity | headache days in a 30 day | ividini vvinidicy C |
| literisity | period from M0 to M2. | |
| | period from 1.10 to 1.12. | |

| Change in Migraine-Specific | Median change in MSQ score | Mann-Whitney U |
|---|---|---|
| Quality of Life – Total, and 3 | from M0 to M2 | |
| subscales | | |
| Change in Hamilton | Median change in Ham-D | Mann-Whitney U |
| Depression Scale | score from M0 to M2 | |
| Tolerability | Side effects | Mann Whitney Us |
| | AEs Total | |
| | AEs related in any degree to | |
| | the treatment | |
| Satisfaction | % of participants who report | Fisher's Exact Test |
| | being satisfied with the | |
| | treatment | |